CLINICAL TRIAL: NCT04433403
Title: A Multicenter Clinical Study on the Detection of Pathogenic Microorganisms in Adult Severe Pneumonia Patients in Liaoning Province
Brief Title: Pathogenic Microorganisms in Adult Severe Pneumonia Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shengjing Hospital (Other)
Collaborators: Chaoyang Central Hospital (Other); Yingkou Central Hospital (Unknown); Huludao central hospital (Unknown); Dandong First Hospital (Unknown); Fushun Mining Bureau General Hospital (Unknown); Benxi Cental Hospital (Other)
Responsible Party: Principal Investigator, Hongyu Zhao, deputy director of emergency department, Shengjing Hospital
Other Study IDs: PMASP
Record Dates: First submitted 2020-06-13; First posted 2020-06-16 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Pathogenic Microorganism of Serious Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pathogenic microorganism — Detection of pathogenic microorganisms in adult severe pneumonia by second generation sequencing

SUMMARY:
This study aimed to evaluate pathogenic microorganisms in adult severe pneumonia patients in different cities of Liaoning Province

DETAILED DESCRIPTION:
The pathogenic microorganisms of adult patients with severe pneumonia is detected in this study. Clinical treatment does not involve , so it meets the ethical requirements. The clinical data, laboratory test results and imaging data of adult severe pneumonia patients in different hospitals in different cities are recorded. The pathogenic microorganism is detected by second-generation sequencing of lower respiratory tract sputum or alveolar lavage fluid samples, and the data were sorted out to draw the pathogenic microorganism spectrum of adult severe pneumonia in Liaoning area. It will be used to guide clinical empirical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the standard of severe pneumonia： Main standards： Requiring mechanical ventilation or septic shock requiring vasoconstrictor therapy.

Secondary standards：(only if 3 items are met) Disturbance of consciousness; respiratory rate ≥ 30 times/min; PaO2/FiO2 ≤ 250, or PaO2 < 60mmHg; azotemia (BUN ≥ 7.12mmol / L); hypotension requires strong fluid resuscitation; infiltration of multiple lobes; leucopenia (WBC < 4 × 109 / L); thrombocytopenia (< 10 × 109 / L); hypothermia (T < 36 ℃).

Exclusion Criteria:

* refuse to sign informed consent; inaccurate results due to unqualified sputum or BALF samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe pneumonia patients, aged 18 years and above, gender unlimited.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathogenic microorganism spectrum of adult severe pneumonia in Liaoning Province | 2020.7-2023.12
  Detection of pathogenic microorganisms in severe pneumonia by second generation sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing hospital of China Medical University, Shenyang, Liaoning, China